CLINICAL TRIAL: NCT01052870
Title: Study Evaluating the Association of CAG Repeat Polymorphisms and Finasteride Response in Women With Androgenetic Alopecia
Brief Title: Association of Polymorphisms in the Androgen Receptor Gene and Finasteride Response in Women With Androgenetic Alopecia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HairDx, LLC (Industry)
Responsible Party: Sharon Keene, M.D., HairDx
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HairDx2009
Record Dates: First submitted 2010-01-16; First posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Androgenetic Alopecia
Keywords: pharmacogenomics, androgen receptor gene, androgen sensitivity, CAG repeats, androgenetic alopecia; Pharmacogenomics in treatment for androgenetic alopecia in women
MeSH Terms: conditions — Alopecia; Bulbo-Spinal Atrophy, X-Linked | interventions — Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- androgen receptor gene polymorphism (Other): Medication response will be assessed according to androgen receptor genotype
  Interventions: Drug: Finasteride
- finasteride (Active Comparator): medication for treating androgenetic alopecia in women
  Interventions: Drug: Finasteride

INTERVENTIONS:
Drug: Finasteride — Effect of 1 mg finasteride on women with androgenetic alopecia depending on their AR gene polymorphism (androgen sensitivity)

SUMMARY:
Previous studies of finasteride treatment in women with hair loss have failed to show positive results, yet, some women have responded anecdotally. Given that polymorphisms of the androgen receptor gene which confer androgen sensitivity impact male response to finasteride therapy, it was hypothesized that the same polymorphism in women may identify the group that will respond. This study is designed to test the impact of finasteride therapy on hair loss in postmenopausal women.

DETAILED DESCRIPTION:
Androgen sensitivity in the cell is determined by the number of Cytosine-Adenine-Guanine repeats in the Androgen Receptor gene. Lower CAG repeats have been associated in previous studies with androgenic conditions such as acne, hirsutism and hair loss in men and women. Keeping this in mind, we tested women with hair loss in the frontal or vertex area, for their AR genotype. Patients were randomized to placebo or 1 mg finasteride therapy for 6 months. Global photographs and 2 tatooed areas of 1cm2 each were measured monthly to assess global appearance and hair counts for medication impact.

ELIGIBILITY:
Inclusion Criteria:

* women with hair loss

Exclusion Criteria:

* pre menopausal,
* metabolic or medication or non-androgenetic causes of hair loss,
* diffuse hair loss

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Keene, M.D., Principal Investigator — HairDx, LLC